CLINICAL TRIAL: NCT01664611
Title: The DREAM Study (Daily Remote Ischaemic Conditioning Following Acute Myocardial Infarction)
Brief Title: Daily REmote Ischaemic Conditioning Following Acute Myocardial Infarction
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); Freemasons' Medical Research Funding (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0306
Record Dates: First submitted 2012-07-19; First posted 2012-08-14 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2012-08

CONDITIONS: Post Myocardial Infarction
Keywords: Remote Ischaemic Conditioning; Remodeling; Heart Failure; Myocardial Infarction; Ischaemia/Reperfusion Injury; successful primary percutaneous coronary intervention following a first STEMI
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Participants in this arm will receive remote ischaemic conditioning on a daily basis for 4 weeks post MI
  Interventions: Procedure: Remote Ischaemic Conditioning administered via the inflation of a blood pressure cuff on the upper arm
- Sham arm (Sham Comparator): Participants in this arm will receive sham ischaemic conditioning on a daily basis for 4 weeks post MI
  Interventions: Procedure: Sham conditioning

INTERVENTIONS:
Procedure: Remote Ischaemic Conditioning administered via the inflation of a blood pressure cuff on the upper arm — Suprasystolic blood pressure cuff inflation for set periods to time to render a limb ischaemic followed by periods of deflation to allow for reperfusion.
  Other Names: The electronic blood pressure cuff used to induce conditioning is the Accoson Greenlight 300.; Cell Aegis AutoRIC machine
  Arms: Treatment arm
Procedure: Sham conditioning — Non therapeutic inflation of a blood pressure cuff that does not cause ischaemia/reperfusion injury
  Arms: Sham arm

SUMMARY:
Remote ischaemic conditioning (RIC) is known to reduce infarct size post MI when used in the peri/immediate post infarct period. However little is known as to the effect of repeated remote conditioning post-MI (Myocardial Infarction) on not only infarct size, but also on ventricular remodeling and ultimately cardiac failure. In this phase II first in man trial, the investigators intend to carry out daily remote ischaemic conditioning in post MI patients. The principal hypothesis is that RIC applied on a daily basis for 4 weeks following a heart attack improves the ejection fraction at 4 months as assessed by cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* LVEF < 45% on baseline ECHO
* First STEMI
* Successful revascularisation by PPCI
* Able to attend regional centre for follow-up appointment
* Competent to consent

Exclusion Criteria:

* < 18 of age
* ICD or CRTP/D in-situ
* Prior history of heart failure
* Haemoglobin < 11.5 g/dl
* Creatinine > 200 µmol/L (eGFR<30ml/min/m2)
* Known malignancy/other comorbid condition which in the opinion of the investigator is likely to have significant negative influence on life expectancy
* Significant complications/illness following MI
* Unable to undergo cMRI
* Further planned coronary interventions
* Enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09-26 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Mean change in LVEF from baseline to 4 months as assessed by cMRI | Participants will be followed for a total of 4 months from date of MI to final outpatient follow-up at which point they will be discharged. Primary outcome measure assessed at baseline and 4 months post MI.
  Mean change in LVEF from baseline to 4 months as assessed by cMRI

SECONDARY OUTCOMES:
Final infarct size at 4 months as assessed by cMRI | Participants will be followed for a total of 4 months from date of MI to final outpatient follow-up at which point they will be discharged. Secondary outcome measure assessed at 4 months post MI.
  Final infarct size at 4 months as assessed by cMRI
Mean blood biomarker levels of heart failure and ventricular remodelling at baseline and 4 months | Participants will be followed for a total of 4 months from date of MI to final outpatient follow-up at which point they will be discharged. Secondary outcome measure assessed at baseline and 4 months post MI.
  Mean blood biomarker levels of heart failure and ventricular remodelling (e.g. NT-proBNP, MMP9, TIMP1) at baseline and 4 months
Mean KCCQ score at 4 months | Participants will be followed for a total of 4 months from date of MI to final outpatient follow-up at which point they will be discharged. Secondary outcome measure assessed at 4 months post MI.
  Mean Kansas City Cardiomyopathy Screen (KCCQ) score at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Samani, FRCP, MD, MBChB, BSc, Principal Investigator — University of Leicester
Locations (1):
- Univesrity of Leicester, Department of Cardiovascular Science, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold JR, P Vanezis A, Rodrigo GC, Lai FY, Kanagala P, Nazir S, Khan JN, Ng L, Chitkara K, Coghlan JG, Hetherington S, Samani NJ, McCann GP. Effects of late, repetitive remote ischaemic conditioning on myocardial strain in patients with acute myocardial infarction. Basic Res Cardiol. 2022 Apr 23;117(1):23. doi: 10.1007/s00395-022-00926-7. PMID 35460434
- [Derived] Vanezis AP, Arnold JR, Rodrigo G, Lai FY, Debiec R, Nazir S, Khan JN, Ng LL, Chitkara K, Coghlan JG, Hetherington SL, McCann GP, Samani NJ. Daily remote ischaemic conditioning following acute myocardial infarction: a randomised controlled trial. Heart. 2018 Dec;104(23):1955-1962. doi: 10.1136/heartjnl-2018-313091. Epub 2018 May 10. PMID 29748420